CLINICAL TRIAL: NCT04134000
Title: Phase Ib Trial of Atezolizumab and BCG in High Risk BCG naïve Non-muscle Invasive Bladder Cancer (NMIBC) Patients: BladderGATE Study
Brief Title: Atezolizumab and BCG in High Risk BCG naïve Non-muscle Invasive Bladder Cancer (NMIBC) Patients (BladderGATE)
Acronym: BladderGATE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion Oncosur (Network)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BladderGATE; 2019-002061-36 (EudraCT Number)
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Invasive Bladder Cancer
Keywords: non-muscle; bladder cancer; näive
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: open-label, non-randomized, dose de-escalation clinical trial with atezolizumab administered by IV infusion in combination with intravesical BCG.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + BCG (Experimental): Ten patient will be enrolled in first cohort, starting on level 0 (DL 0) receiving BCG 1 instillation per week and Atezolizumab 1200 mg IV every three weeks (q3w).
  The next level of dose in case is necessary is BCG 1/2 instillation per week and Atezolizumab 1200 mg IV every three weeks (q3w)
  Interventions: Drug: Atezolizumab; Drug: BCG

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg IV q3w until recurrence of disease, disease progression (e.g., muscle-invasive or metastatic UBC), symptomatic deterioration (i.e., uncontrollable pain secondary to disease or unmanageable ascites, etc.) attributed to disease progression as determined by the investigator, Intolerable toxicity related to atezolizumab, including development of an immune-mediated adverse event determined by the investigator to be unacceptable given the individual patient's potential response to therapy and severity of the event, any medical condition that may jeopardize the patient's safety if he or she continues on study treatment, use of another non-protocol anti-cancer therapy or pregnancy.
Drug: BCG — 1 or 1/2 instillation per week until recurrence of disease, disease progression (e.g., muscle-invasive or metastatic UBC), symptomatic deterioration (i.e., uncontrollable pain secondary to disease or unmanageable ascites, etc.) attributed to disease progression as determined by the investigator, Intolerable toxicity related to atezolizumab, including development of an immune-mediated adverse event determined by the investigator to be unacceptable given the individual patient's potential response to therapy and severity of the event, any medical condition that may jeopardize the patient's safety if he or she continues on study treatment, use of another non-protocol anti-cancer therapy or pregnancy.

SUMMARY:
Patients with high-risk non-muscle invasive bladder cancer (NMIBC) are usually managed by transurethral resection of their bladder tumor (TURBT) alone plus additional intravesical therapy to deliver high local concentrations of a therapeutic agent within the bladder, potentially destroying viable tumor cells that remain following TURBT. Although the exact mechanism of bacillus Calmette-Guerin (BCG) antitumor action is unknown, its intravesical instillation triggers a variety of local immune responses, which appear to correlate with antitumor activity. BCG induction plus maintenance is the current, guideline-recommended standard of care for high-risk NMIBC. Both recent evidence and guidelines suggest that full-dose BCG maintenance after the first BCG dose of induction course as used in the SWOG 8507 and European Organization for Research and Treatment of Cancer (EORTC) 30911 and 30962 trials, is the most appropriate maintenance schedule. High-risk NMIBC patients following adequate treatment have a recurrence rate at 1 and 2 years of 25 and 30% respectively after treatment with the current standard (BCG), which is clearly unsatisfactory. Programmed death ligand 1 (PD-L1) is a surface glycoprotein that functions as an inhibitor of T-cells and plays a crucial role in suppression of cellular immune response. It is implicated in tumor immune escape by inducing apoptosis of activated antigen-specific CD8 T-cells, impairing cytokine production and diminishing the toxicity of activated T-cells. PD-L1 expression by immunohistochemistry using the Ventana SP142 assay on tumor-infiltrating immune cell (IC) status defined by the percentage of PD-L1 positive ICs: IC0 (<1%); IC1 (≥1% but<5%); and IC2/3 (≥5%PD-L1) has been demonstrated to be higher (IC2/3) in resection and TURBT specimens versus biopsies from primary lesions or metastatic sites. In patients with metastatic bladder cancer, treatment with the PD-L1 inhibitor atezolizumab (1200 mg, every 3 weeks) resulted in objective response rates of 26% in the IC2/3 group, 18% in the IC1/2/3 group and 15% in all patients. The median overall survival was 11.4 months in the IC2/3 group, 8.8 months in the IC1/2/3, and 7.9 months in all patients. Grade 3-4 related treatment-related adverse events occurred in 16% and grade 3-4 immune-mediated adverse events occurred in 5% of treated patients. In murine models with invasive bladder cancer, anti-PD-1 plus CpG has shown to increase survival in mice, with anti-PD-1 plus CpG being superior to either agent alone. Taken together, these results confirmed the clinical activity of atezolizumab in metastatic bladder cancer, which could be beneficial in patients with NMIBC in combination with standard approaches such as BCG.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old.
2. Signed Informed Consent Form
3. Histologically confirmed diagnosis of high risk non-muscle-invasive (T1, high grade Ta - G3- and / or carcinoma in situ) transitional cell carcinoma of the bladder
4. Never treated with BCG or stopped >3y ago
5. World Health Organization Performance Status (WHO PS) 0-1
6. No prior radiation to bladder
7. Life expectancy ≥ 5 years
8. Adequate hematologic and end-organ function
9. The time elapsed between the TURBT and the start of the study treatment will not be less than 4 weeks or more than 12 weeks
10. Women who are not postmenopausal or surgically sterile must have a negative serum pregnancy test result within 14 days prior to the first dose of study treatment.
11. For women of childbearing potential: agreement to remain abstinent or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 150 days after the last dose of study drug.
12. Tumor tissue biopsy at study entry or availability of an archival specimen obtained within 2 months of study screening
13. Willingness to complete all study-related procedures including patient-reported questionnaires

Exclusion Criteria:

1. Muscle-invasive, locally advanced non-resectable, or metastatic urothelial carcinoma (i.e., T2, T3, T4, and/or stage IV)
2. Previous BCG within a 3 years period
3. Life expectancy <5 years
4. WHO PS 2, 3 or 4
5. Known additional malignancy that is progressing or requires active treatment
6. Active autoimmune disease that has required systemic treatment in the past 2 years
7. Evidence of interstitial lung disease or active non-infectious pneumonitis
8. Active infection requiring systemic therapy
9. Pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial through 150 days after the last dose of study treatment.
10. Prior therapy with an anti-programmed cell death 1 (PD-1), anti-PD-ligand 2 (L2) agent, or with an agent directed to another co-inhibitory T-cell receptor
11. Known human immunodeficiency virus (HIV)
12. Known active Hepatitis B or C infection or tuberculosis
13. Received a live virus vaccine within 30 days of planned start of study treatment
14. Treatment with any approved anti-cancer therapy, including chemotherapy , radiation therapy , or hormonal therapy within 3 weeks prior to the first dose of study treatment
15. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 4 weeks prior to the first dose of study treatment
16. Allergy or hypersensitivity to components of the atezolizumab or BCG formulation
17. Prior allogeneic stem cell or solid organ transplantation
18. History of idiopathic pulmonary fibrosis, organizing pneumonia , drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
19. Serum albumin < 2.5 g/dL
20. Severe infections within 4 weeks prior to the first dose of study treatment
21. Signs or symptoms of infection within 2 weeks prior to the first dose of study treatment
22. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to the first dose of study treatment
23. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina
24. Major surgical procedure other than for diagnosis within 4 weeks prior to the first dose of study treatment, or anticipation of need for a major surgical procedure during the course of the study
25. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
26. History of prior systemic BCG infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 24 months
  Incidence and nature of DLT of BCG plus atezolizumab combination in NMIBC, graded according to NCI CTCAE v5.
Recurrence free survival. | Up to 24 months
  Time from the date of start of treatment until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from therapy or receives another anticancer therapy prior to progression according to RECIST 1.1 as assessed by the Investigator

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 24 months
  Incidence of Adverse Events (AEs) per patient
Patient reported outcome | Up to 24 months
  The change from baseline in patient-reported symptoms, function, and Health-related quality of life (HRQoL), as measured by the EORTC Quality of Life Questionnaire (QLQ)-C30.
Patient reported outcome | Up to 24 months
  The change from baseline in patient-reported symptoms, function, and HRQoL, as measured by the EORTC Quality of Life Questionnaire (QLQ)-NMIBC24

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Castellano, MD, Principal Investigator — Hospital 12 de Octubre
Locations (1):
- Hospital 12 de Octubre, Madrid, Spain